CLINICAL TRIAL: NCT03508778
Title: CLinical Evaluation of the FluidVision AIOL for Accommodation Restoration
Brief Title: Clinical Evaluation of the FluidVision Accommodation Intraocular Lens (AIOL)
Acronym: CLEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PowerVision (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: CTP08239
Record Dates: First submitted 2018-04-05; First posted 2018-04-26 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Cataract
Keywords: Intraocular lens; Eye surgery
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- FluidVision (Experimental): FluidVision AIOL implanted in the capsular bag of the eye during cataract surgery. Both eyes were implanted, with the second eye surgery occurring after the Week 1 follow up for the first eye surgery.
  Interventions: Device: FluidVision AIOL; Procedure: Cataract surgery
- PanOptix (Active Comparator): Commercially available trifocal IOL implanted in the capsular bag of the eye during cataract surgery. Both eyes were implanted, with the second eye surgery occurring after the Week 1 follow up for the first eye surgery.
  Interventions: Device: AcrySof IQ PanOptix Trifocal IOL; Procedure: Cataract surgery

INTERVENTIONS:
Device: FluidVision AIOL — Investigational implantable medical device intended for long-term use over the lifetime of the cataract subject
  Arms: FluidVision
Device: AcrySof IQ PanOptix Trifocal IOL — Commercially available implantable medical device intended for long-term use over the lifetime of the cataract subject
  Other Names: PanOptix
  Arms: PanOptix
Procedure: Cataract surgery — Cataract surgery per investigator's standard practice

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of an investigational IOL in providing a range of vision as compared to a commercially available trifocal IOL in subjects undergoing cataract extraction and IOL implantation.

DETAILED DESCRIPTION:
Upon obtaining written informed consent and confirmation of subject eligibility via preoperative assessments, subjects were randomized in a 1:1 ratio to receive either the investigational IOL or the commercially available trifocal IOL in both eyes. The second eye for each subject was implanted after completion of the 1-week follow up for the first implanted eye. The expected total duration of participation for each subject was up to 14 months.

ELIGIBILITY:
Key Inclusion Criteria:

* Require cataract extraction by phacoemulsification;
* Corrected Distance Visual Acuity (CDVA) worse than 20/40 Snellen, or presence of visually significant lens opacity;
* Preoperative or predicted postoperative astigmatism of ≤ 1.0 diopter.

Key Exclusion Criteria:

* Use of current medications that may affect accommodation or confound study results;
* Systemic disease that may increase the operative risk or confound results;
* Ocular conditions or degenerative disorders that may predispose the subject to future complications;
* Monocular subjects or significant permanent visual function loss in 1 eye;
* Previous ocular surgery in either eye that may confound the results or increase the risk to the subject.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-02-27 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Distance Corrected Near Visual Acuity (DCNVA) at 100% Contrast - First Implanted Eye | Month 6 postoperative
  Visual acuity was tested at a distance of 40 centimeters with distance correction (plus or minus power) in place.

SECONDARY OUTCOMES:
Distance Corrected Intermediate Visual Acuity (DCIVA) at 100% Contrast - First Implanted Eye | Month 6 postoperative
  Visual acuity was tested at a distance of 66 centimeters with distance correction (plus or minus power) in place.
Distance Corrected Near Visual Acuity (DCNVA) at low contrast - First Implanted Eye | Month 6 postoperative
  Visual acuity was tested at a distance of 40 centimeters with distance correction (plus or minus power) in place.
Percentage of Eyes with 20/32 or Better Visual Acuity Between 4 meters and 40 centimeters on the Defocus Curve | Month 6 postoperative
  A series of plus and minus lenses were placed over the subject's best distance manifest correction to simulate distances from far to hear.

CONTACTS AND LOCATIONS:
Locations (1):
- PowerVision Investigative Site, Somerset West, South Africa

IPD SHARING:
Plan to Share IPD: No